CLINICAL TRIAL: NCT07137468
Title: Excessive Weight, Breast Cancer, and Endocrine Disrupting Chemicals (EDCs): Findings From Active Living After Cancer (ALAC) With Environmental Vitality
Brief Title: Everyday Exposures: How Chemicals and Weight Impact Breast Cancer Risk
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-0698; NCI-2025-06013 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires; Videotape Recording

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-Focus Group Survey: Before your focus group session, you will complete computer-based surveys about your age, biological sex, gender, income, highest level of education, marital status, insurance status, and health behaviors. The online surveys may take up to 40 minutes to complete.
  Interventions: Other: Surveys
- Focus Group Session: After completing the pre-focus group surveys, you will be assigned to a focus group. The focus group will include a warm-up discussion (10 minutes), a short audiovisual presentation (5 minutes) describing endocrine-disrupting chemicals (EDCs), and open-ended questions facilitating discussions on environmental exposures and personal care product usage and ALAC program from your perspective (75 minutes).
  Focus groups will occur by Zoom video conferencing and will be audio- and video-recorded. The recording will be transcribed (written down) word-for-word, but without your name or any other identifying information. The digital audio and video files will be destroyed after they are transcribed.
  Interventions: Other: Video
- Post-Focus Group Survey: After your focus group session, you will complete a computer-based survey to help researchers understand the products you use and things that you do in your everyday life.
  You will also complete a questionnaire asking about the products you've used in the last 24 hours using the Clearya app. The Clearya app captures the ingredients in the products you use by taking pictures or videos of your products. You will be asked to answer 3 questions for each product scanned.
  The online surveys may take up to 40 minutes to complete.
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Electronic surveys will completed via REDCap.
  Groups: Post-Focus Group Survey; Pre-Focus Group Survey
Other: Video — Focus group sessions and community forums will be conducted via videoconference (Zoom)
  Groups: Focus Group Session

SUMMARY:
To learn about breast cancer survivor's knowledge of and interest in learning about environmental exposures related to personal care products. Researchers also want to learn if there is a link between excessive weight and chemicals that may affect hormones.

DETAILED DESCRIPTION:
Primary Objectives:

Excessive body weight, endocrine disrupting chemicals (EDCs), and breast cancer are interconnected through disruptions in hormone balance, with notable disparities in risk and outcomes for under-resourced communities. Excessive weight is a risk factor for breast cancer particularly in postmenopausal individuals, primarily due to increased estrogen production from adipose tissue.

EDCs, such as parabens, bisphenols, and phthalates, have been implicated in both excessive weight and breast cancer, particularly in hormone-sensitive breast cancer subtypes. These non-persistent chemicals are commonly found in personal care products, such as cosmetics and hair care items. Parabens have been shown to promote pro-tumorigenic effects in luminal breast cancer cells, raising concerns about their role in breast cancer incidence. Research has also highlighted that African American individuals face higher exposure to EDCs, especially through hair and other personal care products marketed to people of color, which may contribute to disparities in breast cancer risk.

The relationship between weight and breast cancer is complex with differences in body mass index influencing risk. Under-resourced groups are more likely to be diagnosed with aggressive late-stage breast cancer, a risk further exacerbated by high body weight. Moreover, disparities in healthcare access, economic and social standing, and exposure to EDCs, also known as non-medical drivers of health (NMDOH), may compound breast cancer mortality rates in these communities.

The overall goal of this proposal is to engage participants from the ALAC program and determine their knowledge and interest in environmental exposure education focused on personal care products. The information gained from our efforts will support the development of the Active Living After Cancer with Environmental Vitality (ALAC-ENV) intervention to improve QOL.

Additionally, we will determine the association between prevalent EDCs and excessive weight for breast cancer survivors. To achieve this goal, we will pursue the following specific aims:

Specific Aim 1: Determine breast cancer survivors' environmental exposure knowledge. Participants (n=30; pilot-tested group (n=6-8)) will participate in focus group interviews to assess their interest and understanding of environmental exposures with an emphasis on personal care products. Participants in the pilot-testing group will assist with potential modifications regarding the focus group guide. Participants in the pilot-testing group will be recognized as "Focus Group 1" participants and will complete all protocol procedures.

Specific Aim 2: Determine the relationship between exposures to prevalent EDCs and BMI. A cross-sectional design to examine associations between BMI and measurements of non-persistent EDCs in urine samples of cancer survivors.

Emerging evidence on the disproportionate exposure to carcinogenic chemicals and its role in cancer-related disparities underscores the need for this study. The limited understanding of the relationship between EDCs and weight-related cancers further highlights the importance of exploring pathways to mitigate health risks in under-resourced communities. Findings from this study will inform an R-level grant to develop a randomized trial testing the efficacy of an adapted ALAC-ENV curriculum for dissemination and implementation in community settings. Additionally, we will seek foundation grant support for a cross-sectional study examining the association between body mass index, EDC exposure, and cancer in Acres Homes within the context of NMDOH.

ELIGIBILITY:
Inclusion Criteria:

1. Be a resident of Acres Home community
2. Be 18 years of age and older
3. Current or former participants of the ALAC program
4. Self-report a breast cancer diagnosis including subtypes
5. Able to communicate in English

Exclusion Criteria:

1. Self-report metastatic breast cancer diagnosis
2. Unable to communicate in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: MD Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcome Measure | Through study completion; an average of 1 year
  Questionnaires/Videos

CONTACTS AND LOCATIONS:
Overall Officials: Dede Teteh-Brooks, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org